CLINICAL TRIAL: NCT02457520
Title: An Open-label Study Evaluating the Long-term Efficacy, Quality of Life, and Safety of ABSORICA® (Isotretinoin) Capsules Administered Without Food in Patients With Severe Recalcitrant Nodular Acne
Brief Title: ABSORICA in Patients With Severe Recalcitrant Nodular Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABS157LT
Record Dates: First submitted 2015-05-16; First posted 2015-05-29 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single treatment arm (Experimental): ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
  Other Names: ABSORICA

SUMMARY:
This is an uncontrolled, open-label study being conducted in approximately 200 healthy males, non-pregnant, non-nursing females, age 12 to 45 years, with severe recalcitrant nodular acne.

ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day will be administered for 4 weeks followed by 1.0 mg/kg/day for 16 weeks. Female subjects consenting to use two forms of birth control or abstinence are included.

DETAILED DESCRIPTION:
This study is designed to collect efficacy, safety, and quality of life (QOL) data from subjects who receive Absorica® without food. The study will investigate the treatment efficacy, frequency of relapse once the treatment has been discontinued, quality of life during the active treatment and during a 2-year post treatment period and the overall safety of treatment with Absorica®.

This is a single-arm, open-label study consisting of 2 phases: a 20-week (5-month) open-label Active Treatment Period (ATP) and a 104-week (2-year) post treatment period (PTP). The total study duration is to be 124 weeks, excluding a screening period. During the ATP, after week 2 visit, visits will be scheduled at 4-week intervals for a total of 8 visits (1 screening visit, 1 baseline visit, and 6 on-study visits). During the PTP, the first visit will be 4 weeks after End of Treatment (EOT), the second visit will be 12 weeks after EOT, and subsequent visits will be scheduled at 26-week (± 2 weeks) intervals for a total of 6 visits.

ELIGIBILITY:
General Inclusion Criteria Subjects must meet the following mandatory inclusion criteria at the time of screening to be eligible to enter the study and must agree to conform to the requirements of the study and the iPLEDGE program.

* Written informed consent, including mandatory photographic consent, on a gender-specific informed consent form (ICF) & Health Insurance Portability and Accountability Act (HIPAA) authorization prior to the performance of any study-related procedures.
* Pregnant females and females who are not to become pregnant during the ATP phase of the trial and for 30 days after receiving their last dose of study drug.
* Female subjects of childbearing potential ready to use 2 forms of effective contraception simultaneously for 1 month before starting Absorica® (isotretinoin), while taking Absorica® & for 1 month after Absorica® has been stopped.
* Male and female subjects of non-childbearing potential

Specific Inclusion Criteria:

* Severe recalcitrant nodular acne.
* Five or more nodule lesions on the face.
* Treatment-naïve subjects.
* Age between 12 and 45 years.
* Weight between 40 and 110 kg.
* Female subjects of childbearing potential only: Negative results from serum pregnancy tests with a sensitivity of at least 25 milli-international unit/mL.
* Good general health as determined by the investigator based on the subject's medical history, physical examination, vital signs measurements, and laboratory test results.
* Subjects who present with stable & controlled diabetes mellitus (Types I and II).
* Subjects with previously diagnosed polycystic ovarian syndrome (PCOS) can be included in the study if in the opinion of the investigator they do not have any other clinically significant abnormality (eg, metabolic syndrome or elevated lipids

Exclusion Criteria:

General Exclusion Criteria

* Presence of any clinically significant physical examination finding, vital signs measurement, or abnormal laboratory value;
* Presence of a beard or other facial hair that could interfere with the study assessments;
* Participated in another clinical trial or received an investigational product within 3 months prior to screening;
* History of excessive or suspected abuse of alcohol (based on the clinical judgment of the investigator), recreational drugs, and/or drugs of abuse, e.g., club drugs, cocaine, ecstasy/ methylenedioxymethamphetamine, heroin, inhalants, marijuana, methamphetamine, phencyclidine, prescription medications, anabolic steroids, etc.
* Use of prohibited or restricted prior or concomitant medications. Female Specific Exclusion Criteria
* Are pregnant;
* Are at a high risk for becoming pregnant or likely to become pregnant during treatment;
* Are breast-feeding or considering breast-feeding during the course of the study;
* Have a known history of PCOS with another clinically significant abnormality (eg, metabolic syndrome or elevated lipids);
* Are unable or unwilling to maintain compliance with birth control measures

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 201 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Anvekar, MD, Study Director — Ranbaxy Laboratories Limited
Locations (1):
- Texas Dermatology and Laser Specialists, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Rosso JQ, Stein Gold L, Segal J, Zaenglein AL. An Open-label, Phase IV Study Evaluating Lidose-isotretinoin Administered without Food in Patients with Severe Recalcitrant Nodular Acne: Low Relapse Rates Observed Over the 104-week Post-treatment Period. J Clin Aesthet Dermatol. 2019 Nov;12(11):13-18. Epub 2019 Nov 1. PMID 32038751

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Treatment Arm: Absorica capsules 0.5 mg/kg/day for 4 weeks, followed by 1.0 mg/kg/day for 16 weeks.
Period: Active Treatment Phase
Arm/Group | Single Treatment Arm
Started | 201 (All subjects received treatment according to the same regimen.)
Completed (Subjects Completing Treatment Phase, n (%)) | 167
Not Completed | 34
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 8
Not completed — Non-compliance with Study Treatment | 3
Not completed — other | 4
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Period: Post-treatment Period
Arm/Group | Single Treatment Arm
Started | 167
Completed | 119
Not Completed | 48
Not completed — Other: Retreatment Required | 7
Not completed — Lost to Follow-up | 23
Not completed — Other | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Population: safety population
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 170
  Unknown or Not Reported | NA — Only Hispanic or Latino and Non-Hispanic or Latino were included in the study
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 167
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 201

OUTCOME MEASURES:

1. Primary Outcome: Active Treatment Period: Total Acne-Specific Quality of Life Score at Week 20
Description: There are 4 domains: self-perception (22 questions), role-social (50 questions), role-emotional (33 questions), and acne symptoms (85 questions) in the acne-QOL questionnaires.
  Calculation of the domain scores was accomplished by summing all item responses within each domain.
  Self-perception: The range of possible scores is 0 to 30 points. Role-social: The range of possible scores is 0 to 24 points. Role emotional: The domain scores range from 0 to 30 points. Acne symptoms: The domain scores range from 0 to 30 points.
Time Frame: Week 20
Population: This endpoint was analyzed in the per-protocol population and the number of participants analyzed in the per-protocol population set was 166.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 166
score | 100.7 (18.1)

2. Primary Outcome: Primary Efficacy Endpoint, Post-treatment Period: Subjects Requiring Retreatment During the Post-treatment Period and Time to Retreatment
Description: subjects who were at least 75% compliant with their assigned treatment, had no major protocol violations, had a Week 20 count of total nodular lesions, and did not use any disallowed medications during the 20 weeks of treatment. (Retreated with Oral Isotretinoin Per Protocol Population).
Time Frame: 20 weeks
Population: Per Protocol Population
Measure: Number; unit: number of subjects
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 163
number of subjects | 7

3. Secondary Outcome: Active Treatment Period- Change From Baseline in Lesion Counts at Week 20
Description: Change from baseline in the lesion count (nodules and inflammatory lesions) at the end of the ATP. (Per Protocol Population)
Time Frame: Baseline and at week 20
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 166
percentage change in lesion count | -89.14 (16.36)

4. Secondary Outcome: Active Treatment Period-Change From Baseline in Acne-Specific Quality of Life Total Score at Weeks 4, 8, 12, and 16
Description: as for outcome 1
Time Frame: Baseline, at week 4, week 8, week 12, and week16
Population: PP population
Measure: Mean (Standard Deviation); unit: score
Groups:
- Single Treatment Arm-Week 16: Visit 7/Week 16
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
- Single Treatment Arm-Week 12: Visit 6/Week 12
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
- Single Treatment Arm-Week 8: Visit 5/Week 8
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
- Single Treatment Arm-Week 4: Visit 4/Week 4
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm-Week 16 | Single Treatment Arm-Week 12 | Single Treatment Arm-Week 8 | Single Treatment Arm-Week 4
Number analyzed (Participants) | 159 | 163 | 162 | 149
score | 32.7 (28.1) | 26.3 (24.6) | 17.8 (22.4) | 14.5 (19.6)

5. Secondary Outcome: Active Treatment Period- Investigator's Global Assessment at Week 20
Description: Investigator's Global Assessment score:
  0 = Clear
  1. = Almost Clear
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very Severe
Time Frame: week 20
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 166
score | -3.1 (1.1)

6. Secondary Outcome: Active Treatment Period- Change From Baseline in Acne-Specific Quality of Life Domain Scores by Domain at Weeks 4, 8, 12, and 16
Description: Acne-Specific Quality of Life, by domain:
  Self Perception: response on 0- to 6-point scale; the range of possible scores is 0 to 30 points.
  Role-social: response on 0- to 6-point scale; the range of possible scores is 0 to 24 points.
  Role-emotional: response on 0- to 6-point scale, exactly the same as those used for the Self Perception and Role-social domains.
  Acne Symptoms:response on 0- to 6-point scale, domain scores range from 0 to 30 points
Time Frame: 20 weeks
Population: per protocol population
Measure: Mean (Standard Deviation); unit: score
Groups:
- Single Treatment Arm-Self Perception; Single Treatment Arm-Role-Emotional; Single Treatment Arm-Role-Social; Single Treatment Arm-Acne Symptoms: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm-Self Perception | Single Treatment Arm-Role-Emotional | Single Treatment Arm-Role-Social | Single Treatment Arm-Acne Symptoms
Number analyzed (Participants) | 166 | 166 | 166 | 166
score
  Visit 8/Week 20 | 10.6 (8.9) | 10.5 (8.7) | 6.5 (7.1) | 11.6 (6.1)
  Visit 7/Week 16: number analyzed (Participants) | 159 | 159 | 159 | 159
  Visit 7/Week 16 | 8.8 (8.8) | 8.7 (8.7) | 5.4 (7.1) | 9.7 (6.2)
  Visit 6/Week 12: number analyzed (Participants) | 163 | 163 | 163 | 163
  Visit 6/Week 12 | 7.0 (7.9) | 6.9 (7.8) | 4.3 (6.0) | 8.2 (5.9)
  Visit 5/Week 8: number analyzed (Participants) | 162 | 162 | 162 | 162
  Visit 5/Week 8 | 4.6 (7.1) | 4.5 (7.1) | 2.6 (5.3) | 6.1 (5.6)
  Visit 4/Week 4: number analyzed (Participants) | 149 | 149 | 149 | 149
  Visit 4/Week 4 | 3.6 (6.3) | 4.0 (6.5) | 2.1 (5.2) | 4.8 (5.0)

7. Secondary Outcome: Active Treatment Period- Change From Baseline in Nodule Count at Week 20
Time Frame: Baseline, and at week20
Measure: Mean (Standard Deviation); unit: percentage change in nodule count
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 166
percentage change in nodule count | -96.18 (11.42)

8. Secondary Outcome: Post-treatment Period- Proportion of Subjects Requiring Treatment With Anti-Acne Medication and Time to Retreatment
Description: Retreated with Prescription Anti-Acne Medication, n/Na (%); Over-the-Counter Anti-Acne Medication and Prescription or Over-the-Counter Anti-Acne Medication- Per Protocol Population.
Time Frame: 104 weeks
Population: PP population
Measure: Count of Participants; unit: Participants
Groups:
- Single Treatment Arm-Retreat With Prescription Anti-acne Medic; Single Treatment Arm - Retreat With Over-the-counter Anti-acne; Single Treatment Arm- Retreat With Prescription or Over-the-co: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm-Retreat With Prescription Anti-acne Medic | Single Treatment Arm - Retreat With Over-the-counter Anti-acne | Single Treatment Arm- Retreat With Prescription or Over-the-co
Number analyzed (Participants) | 163 | 163 | 163
Participants | 22 | 8 | 25

9. Secondary Outcome: Post-treatment Period- Severity of Acne by Lesion Count at Time of Retreatment With Oral Isotretinoin
Description: change from Baseline
Time Frame: 104 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Groups:
- Single Treatment Arm- Total; Single Treatment Arm -Non-inflammatory; Single Treatment Arm-Inflammatory: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm- Total | Single Treatment Arm -Non-inflammatory | Single Treatment Arm-Inflammatory
Number analyzed (Participants) | 7 | 7 | 7
percentage change in lesion count | -20.81 (31.15) | -1.41 (95.81) | -31.53 (19.78)

10. Secondary Outcome: Post-treatment Period- Severity of Acne by Investigator's Global Assessment at Time of Retreatment With Oral Isotretinoin
Description: as for outcome 5
Time Frame: 104 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
score | 3.0 (0.6)

11. Secondary Outcome: Post-treatment Period- Severity of Acne by Lesion Count at Time of Retreatment With Prescription Other Than Oral Isotretinoin
Description: Change from baseline
Time Frame: 104 weeks
Population: (Per Protocol Population)
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Groups:
- Single Treatment Arm-Inflammatory; Single Treatment Arm -Non-inflammatory; Single Treatment Arm- Total: Change from baseline
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm-Inflammatory | Single Treatment Arm -Non-inflammatory | Single Treatment Arm- Total
Number analyzed (Participants) | 22 | 22 | 22
percentage change in lesion count | -66.16 (25.93) | -72.90 (30.52) | -69.83 (22.48)

12. Secondary Outcome: Post-treatment Period- Severity of Acne by Investigator's Global Assessment Score at Time of Retreatment With Over-the-Counter Medication
Description: as for outcome 5
Time Frame: 20 weeks
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 8
score | 1.8 (0.7)

13. Secondary Outcome: Post-treatment Period-Severity of Acne by Lesion Count at Each Visit During the Post-treatment Period
Time Frame: week 124
Population: PP Population
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Arm/Group | Single Treatment Arm-Inflammatory | Single Treatment Arm -Non-inflammatory | Single Treatment Arm- Total
Number analyzed (Participants) | 118 | 118 | 118
percentage change in lesion count | -86.85 (18.89) | -80.45 (37.10) | -85.35 (21.65)

14. Secondary Outcome: Post Treatment Period- Severity of Acne by Nodule Count at Each Visit During the Post-treatment Period
Description: Change from Baseline-Week 124
Time Frame: week 124
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 118
percentage change in lesion count | -99.03 (5.13)

15. Secondary Outcome: Severity of Acne by Investigator's Global Assessment Score at Each Visit During the Post-treatment Period
Description: as for outcome 5
Time Frame: week 124
Population: per protocol population
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 118
score | -3.1 (1.0)

16. Secondary Outcome: Post-treatment Period- Severity of Acne by Lesion Count at Time of Retreatment With Over-the-Counter Medications
Description: Change from Baseline
Time Frame: 20 weeks
Population: (Per Protocol Population)
Measure: Mean (Standard Deviation); unit: percentage change in lesion count
Arm/Group | Single Treatment Arm-Inflammatory | Single Treatment Arm -Non-inflammatory | Single Treatment Arm- Total
Number analyzed (Participants) | 8 | 8 | 8
percentage change in lesion count | -66.61 (17.26) | -63.70 (38.38) | -67.04 (21.87)

17. Secondary Outcome: Post Treatment Period-Severity of Acne by Investigator's Global Assessment Score at Time of Retreatment With Prescription Other Than Oral Isotretinoin
Description: as for outcome 5
Time Frame: 20 weeks
Population: (Per Protocol Population)
Measure: Mean (Standard Deviation); unit: score
Groups:
- Single Treatment Arm: Change from Baseline
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 22
score | -2.4 (1.0)

18. Other Pre Specified Outcome: Post Treatment Period- Acne-Specific Quality of Life by Total Scores at the End of the Post-treatment Period
Description: as for outcome 1
Time Frame: Visit 14/Week 124
Population: PP Population
Measure: Mean (Standard Deviation); unit: score
Groups:
- Single Treatment Arm- Visit 14/ Week 124: Change from Baseline
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
Arm/Group | Single Treatment Arm- Visit 14/ Week 124
Number analyzed (Participants) | 118
score | 44.4 (29.3)

19. Other Pre Specified Outcome: Post-treatment Period- Acne-Specific Quality of Life by Domain Scores at the End of the Post-treatment Period
Description: Acne-Specific Quality of Life, total and by domain:
  Self Perception: response on 0- to 6-point scale; the range of possible scores is 0 to 30 points.
  Role-social: response on 0- to 6-point scale; the range of possible scores is 0 to 24 points.
  Role-emotional: response on 0- to 6-point scale, exactly the same as those used for the Self Perception and Role-social domains.
  Acne Symptoms:response on 0- to 6-point scale, domain scores range from 0 to 30 points
Time Frame: Visit 14/Week 124
Population: per protocol population
Measure: Mean (Standard Deviation); unit: score
Groups:
- Single Treatment Arm-Self Perception; Single Treatment Arm-Role-Emotional; Single Treatment Arm-Role-Social: Change from Baseline
  ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks.
  Isotretinoin: ABSORICA® (isotretinoin) capsules 0.5 mg/kg/day for 4 weeks followed by 1.0 mg/kg/day for 16 weeks
- Single Treatment Arm-Acne Symptoms: Change from Baseline
Arm/Group | Single Treatment Arm-Self Perception | Single Treatment Arm-Role-Emotional | Single Treatment Arm-Role-Social | Single Treatment Arm-Acne Symptoms
Number analyzed (Participants) | 118 | 118 | 118 | 118
score | 12.5 (8.8) | 12.6 (9.1) | 7.7 (7.5) | 11.5 (6.6)

ADVERSE EVENTS:
Time Frame: Active Treatment Period- 20 weeks Post-treatment Period- 124 weeks
Description: All safety analyses were carried out using the safety population, which was defined as all subjects who received at least 1 dose of study treatment. Thus, overall results are depicted for all the subjects
Groups:
- Single Treatment Arm: Absorica capsules 0.5 mg/kg/day for 4 weeks, followed by 1.0 mg/kg/day for 16 weeks.
  Study ABS1517LT was a Phase 4, open-label, single-arm study in subjects with severe recalcitrant nodular acne, consisting of 2 phases: a 20-week (5-month) Active Treatment Phase and a 104-week (2-year) Post Treatment Period.
Arm/Group | Single Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/201
Serious Adverse Events (participants affected / at risk) | 1/201
Other Adverse Events (participants affected / at risk) | 54/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Treatment Arm (N=201)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Treatment Arm (N=201)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (23)
Lip dry (Gastrointestinal disorders) | 23 (23)
Depression (Psychiatric disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02457520/Prot_SAP_000.pdf